CLINICAL TRIAL: NCT01369459
Title: Family-Based Protocol for Medication Integration in Treatment of Comorbid ASU/ADHD
Brief Title: Medication Integration in Treatment of Comorbid Adolescent Substance Users/Attention Deficit Hyperactivity Disorder
Acronym: MIP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The National Center on Addiction and Substance Abuse at Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Aaron Hogue, Director of Adolescent & Family Research, The National Center on Addiction and Substance Abuse at Columbia University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASA2011MIP; 1R21DA031305-01A1 (NIH)
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Attention Deficit Hyperactivity Disorder; Attention Deficit Disorder
Keywords: Comorbid; ADHD; SUD; ASU
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — MIP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Counseling with MIP Protocol (Experimental): We intend for MIP to be a 5-session, family-based protocol delivered during the early portion of ASU treatment. MIP will contain three elements deemed essential for integrating pharmacological interventions into outpatient behavioral treatment for youth: (1) standardized psychiatric assessment and family-focused psychoeducation about the target problem; (2) an approved medication regimen with demonstrated efficacy for comorbid populations; (3) family-based interventions for medication acceptance and coordination of psychiatric and behavioral services. MIP will incorporate research-proven interventions from each of these core areas.
  Interventions: Behavioral: MIP Protocol
- Historical Control (No Intervention)

INTERVENTIONS:
Behavioral: MIP Protocol — We intend for MIP to be a 5-session, family-based protocol delivered during the early portion of ASU treatment. MIP will contain three elements deemed essential for integrating pharmacological interventions into outpatient behavioral treatment for youth: (1) standardized psychiatric assessment and family-focused psychoeducation about the target problem; (2) an approved medication regimen with demonstrated efficacy for comorbid populations; (3) family-based interventions for medication acceptance and coordination of psychiatric and behavioral services. MIP will incorporate research-proven interventions from each of these core areas.
  Arms: Family Counseling with MIP Protocol

SUMMARY:
The goal of this project is to develop and test a brief protocol designed to systematically integrate pharmacological interventions for Attention Deficit Hyperactivity Disorder (ADHD) into behavioral treatment services for adolescent substance users with co-morbid ADHD in everyday care. Primary study aims will yield proof-of-concept data on MIP feasibility and fidelity in usual care and evidence of MIP impact on psychiatric and behavioral services utilization, medication acceptance and compliance, and satisfaction with treatment services.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17 years
* Caregiver able to participate in treatment
* One day of alcohol use to intoxication or illegal drug use in the past 30 days (or 30 days prior to living in a controlled environment)
* endorsement of one or more DSM-IV symptoms of Substance Use or Alcohol Dependence/Abuse
* meet ASAM criteria for outpatient substance use treatment
* meet DSM-IV criteria for ADHD (with or without onset prior to age 7)
* not enrolled in any behavioral treatment

Exclusion Criteria:

* MDD
* Bipolar Disorder
* Mental Retardation
* PDD
* medical or psychiatric illness requiring hospitalization
* current psychotic features
* currently suicidal

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Mini International Neuropsychiatric Interview (MINI) Version 5.0 | Follow-up in 3 months
  MINI is a structured diagnostic interview that assesses DSM-IV diagnoses in adolescents and is designed for administration by lay interviewers. Adolescents and caregivers will complete the Inattentive and Hyperactive/Impulsive scales.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function (BRIEF) | Follow-up at 3-months
  The BRIEF is a parent-report measure of behavioral problems linked to executive functioning and commonly observed in ADHD youth. The BRIEF has been validated on ADHD outpatient samples and teens with mixed clinical diagnoses. This study will use 4 scales: Inhibition, Behavioral Shift, Emotional Control, Plan/Organize.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron T Hogue, Ph.D., Principal Investigator — The National Center on Addiction and Substance Abuse at Columbia University
Locations (1):
- Roberto Clemente Center, New York, New York, United States